CLINICAL TRIAL: NCT06480175
Title: Comparative Study Between Cervical Medial Branch Radiofrequency Ablation Versus Radiofrequency Plus Superficial Cervical Plexus Block in Treatment of the Cervical Facet and Cervical Spondylosis Pain
Brief Title: Radiofrequency Plus Superficial Cervical Plexus Block in Treatment of Cervical Spondylosis Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Lydia edward aziz zakhary, lecturer, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: neck pain
Record Dates: First submitted 2024-06-17; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Neck Pain; Cervical Spondylosis
MeSH Terms: conditions — Neck Pain; Spondylosis | interventions — Cervical Plexus Block; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cervical plexus block (Experimental): patients will receive cervical radiofrequency nerve ablation on both sides and after 2 weeks will be readmitted and will receive superficail cervical plexus block on only one side
  Interventions: Procedure: cervical plexus block

INTERVENTIONS:
Procedure: cervical plexus block — patients will receive cervical radiofrequency ablation on both sides then after 2 weeks they will be readmitted and will receive superficial cervical plexus block on one side only
  Other Names: radiofrequency ablation

SUMMARY:
The goal of this clinical trial is to compare the effectiveness in the pain relief between doing radiofrequency ablation for the medial branch of the cervical facet pain alone vs using it combined with superficial cervical plexus block.in adults patients with cervical spondylosis pain

The main question it aims to answer is:

does adding superficial cervical plexus block to radiofrequency in patients with chronic neck pain provide better analgesia than radioprequency alone ?

DETAILED DESCRIPTION:
participants will be placed in prone position with neck preparation using an iodine-based product and drape in a sterile manner Then the ground pad of the radiofrequency machine will be placed on the back ( the Neurotherm NT1100 regenerator will be used) All the patients will be monitored by ECG, noninvasive blood pressure and pulse oximetry.

The entry sites will be detected under fluoroscopy then local anesthesia will be performed using lidocaine 2% followed by the insertion of the radiofrequency cannula (STRYKER 20 G, 9 cm with 1 cm active tip) targeting the medial branches supplying C4, C5, C6 & C7 bilateral.

the investigators will use 1 entry site for each side and then redirect the needles .

Confirmation of the appropriate location will be done on fluoroscopy in both A-P and lateral views Once targeted, sensory stimulation will be done and every patient is asked if he feels the same pain as that he used to suffer from. Once confirmed with absence of motor response; 1 more ml of lidocaine 20 % is injected and then start our ablation for 180 sec at 80 degrees

The procedure will be done bilateral the same. After 2 weeks , patient will be readmitted and then the investigators will choose to inject the superficial cervical plexus with 5 ml of lidocaine 20% plus 40 mg triamcinolone. injection was random in the right or left side using ultrasound to confirm success.

The side of the block will be recorded for each patient either right or left. Comparison will be done between both sides to study the effect of adding superficial plexus block to radio-frequency whether the analgesic effect is better on the side of radio frequency alone or the side where the superficial cervical plexus block was added to radio-frequency.

The patients will then be asked to be followed up after 1 month and after 6 months and about the improvement in the numeric pain score (NPS) and the patient global impression of change (PGIC) and if they feel that one side is better than the other or they feel the same. Visual analogue score scale will be recorded for documentation.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Age between 30-70 years.
* American society of anesthesiologist ASA 1,2 & 3 physical status.
* MRI cervical spine diagnosing cervical facet arthropathy originating pain .
* Failed full dose medical treatment and life style modification and physiotherapy for 3 months prior to intervention.

Exclusion Criteria:

* Neurological disorders.(previous central and peripheral CNS affection ).
* coagulopathy INR > 1.8 or platelets < 50,000.
* Infection at or near the injection site.
* Presence of pacemaker or defibrillator.
* known allergy to used medications.
* age >70 or <30 years.
* patients with previous history of Radiotherapy , chemotherapy or metastasis
* pregnant patients.
* patients with rheumatological disorders ( rheumatoid arthritis, diffuse idiopathic skeletal hyerostosis, psoriatic arthritis, spondyloarthritis)
* patients with antiphospholipid syndtrome.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
pain releif | 1 months
  evaluating degree of pain releif after cervical medial branch radiofrequency ablation Monitoring pain score using numeric pain rating scale (NPRS) it is a 11 point scale scored from 0-10
  * 0 represents no pain
  * 10 represents the worst pain imaginable . versus radiofrequency plus superficial cervical plexus block by using numeric pain rating scale after 1 month

SECONDARY OUTCOMES:
improved life style | 6 months
  Secondary outcomes that will be detected in our study is the degree of pain releif after 6 months Monitoring pain score using numeric pain rating scale (NPRS) it is a 11 point scale scored from 0-10
  * 0 represents no pain
  * 10 represents the worst pain imaginable .
    * change the need for the use of oral or parentral analgesics
global impression of change | 6 months
  measuring patient global impression of change ( PGIC) score: PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." where score 1 indicating " very much improved " and 7 indicating " very much worse".

CONTACTS AND LOCATIONS:
Overall Officials: lydia zakhary, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

REFERENCES:
- [Background] Berger AA, Liu Y, Mosel L, Champagne KA, Ruoff MT, Cornett EM, Kaye AD, Imani F, Shakeri A, Varrassi G, Viswanath O, Urits I. Efficacy of Dry Needling and Acupuncture in the Treatment of Neck Pain. Anesth Pain Med. 2021 Apr 3;11(2):e113627. doi: 10.5812/aapm.113627. eCollection 2021 Apr. PMID 34336626
- [Background] Burnham T, Conger A, Salazar F, Petersen R, Kendall R, Cunningham S, Teramoto M, McCormick ZL. The Effectiveness of Cervical Medial Branch Radiofrequency Ablation for Chronic Facet Joint Syndrome in Patients Selected by a Practical Medial Branch Block Paradigm. Pain Med. 2020 Oct 1;21(10):2071-2076. doi: 10.1093/pm/pnz358. PMID 32022889